CLINICAL TRIAL: NCT04324320
Title: Psychological Distress in Outpatient Oncological Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Richard Crevenna, Univ. Prof. Dr., MBA, MMSc, Head of the Department of Physical Medicine, Rehabilitation and Occupational Medicine, Medical University of Vienna
Other Study IDs: 1162/2020
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Distress; Oncology
Keywords: outpatient oncological rehabilitation; psychological distress; cross-sectional study
MeSH Terms: conditions — Neoplasms | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- outpatients (oncological rehabilitation): the population studied in this cross-sectional study includes patients with malignant tumour diseases and benign CNS tumours who present to the Outpatient Clinic for Oncological Rehabilitation at the Department of Physical Medicine and Rehabilitation of the Medical University of Vienna
  Interventions: Diagnostic Test: medical assessment; Diagnostic Test: psychological assessment

INTERVENTIONS:
Diagnostic Test: medical assessment — medical assessment includes the collection of
  * sociodemographic data
  * anthropometric data (weight, height, body mass index)
  * medical data
  * psycho-oncologic basis assessment (PO-BADO questionnaire)
  * pain assessment (VAS: visual analogue scale)
  * 3 functional tests:
    * handgrip strength
    * 6 Minute Walking Test
    * Timed Get up and Go Test
Diagnostic Test: psychological assessment — psychological assessment includes several standardized screening and assessment questionnaires and tools:
  * quality of life: SF-36
  * anxiety, depression, stress: Hospital Anxiety and Depression Scale (HADS-D)
  * subjective stress perception: Perceived Stress Scale (PSS-10)
  * resilience: resilience scale (RS-13)
  * fatigue: Brief Fatigue Inventory (BFI)
  * disability related to pain: Pain Disability Index (PDI)
  * workability: Work Ability Index - short version (WAI-K)
  * psychological assessment based on the checklist of the International Diagnoses (IDCL) for ICD-10 and the ICD-10 checklist of symptoms for psychological disorders (SCL))

SUMMARY:
The aim of the study is to assess psychological distress and co-morbidity as well as relevant sociodemographic, anthropometric, medical and functional data in patients treated at the Outpatient Clinic for Oncological Rehabilitation at the Department of Physical Medicine, Rehabilitation and Occupational Medicine at the Medical University of Vienna.

DETAILED DESCRIPTION:
Psychological distress in cancer patients is higher than in the average population and is associated with a lower health-related quality of life. In the course of the disease and its treatment, a psychological distress reaction can lead to a psychosocial crisis and a mental disorder that requires treatment. On average, 25% of all cancer patients suffer from depression, anxiety or adjustment disorders at any point in the course of their disease, and an average of 32% of all cancer patients express the need for psychosocial support. With an increasing reduction in inpatient length of stay times, outpatient care gains growing importance in the context of psycho-oncological diagnostics and aftercare. The overlap between physical symptoms due to cancer diagnosis and treatment and physical symptoms that are related to psychological burdens requires sensitive psycho-oncological diagnostics. This should be carried out as early as possible in the course of the disease so that existing psychological distress can be recognized early and thus a progression of the symptoms can be prevented.

The study aims to assess psychological distress and co-morbidity as well as relevant sociodemographic, anthropometric, medical and functional data in patients treated at the Outpatient Clinic for Oncological Rehabilitation at the Department of Physical Medicine, Rehabilitation and Occupational Medicine at the Medical University of Vienna.

Results should serve as a basis for further individual treatment recommendations.

By ascertaining the psychological distress, appropriate support and treatment measures can be recommended to the patients at an early stage, which help to improve the symptoms, enable participation and thus improve the quality of life of the patients. The assessment of the current individual need for psychological care also helps to refer patients to an inpatient oncological rehabilitation setting that provides the care that is needed more appropriately.

Results should also improve the psychological care of oncologic patients in general. Based on the findings, the psychological care offered within the framework of the current outpatient and inpatient oncological rehabilitation setting could be adapted and expanded as necessary. The results of the study should serve to integrate psycho-oncological care into the overall outpatient oncological rehabilitation concept.

A monocentric cross-sectional study is to be carried out on 165 patients with malignant tumour diseases as well as benign central nervous system tumours over a period of approximately 2 years.

Medical assessment of sociodemographic, anthropometric, medical and functional data will be performed. The gained information is also relevant for physical therapy prescription and treatment recommendations given by the physiatrist at the outpatient clinic for oncological rehabilitation.

Psychological distress and the need for psycho-oncological care for outpatients is determined through standardized screening and suitable assessment procedures. Patients will receive an immediate therapy recommendation regarding their psychological complaints by the clinical psychologist and psychotherapist who performs the assessment.

ELIGIBILITY:
Inclusion Criteria:

* patients with malignant tumour diseases and benign CNS tumours who present to the Outpatient Clinic for Oncological Rehabilitation at the Department of Physical Medicine, Rehabilitation and Occupational Medicine at the Medical University of Vienna
* patients who agree to participate in the study

Exclusion Criteria:

* bad physical condition that does not enable the patient to participate in the study
* language barriers (insufficient understanding of the German language)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with all kinds of malignant tumour diseases and benign CNS tumours who present to the Outpatient Clinic for Oncological Rehabilitation at the Department of Physical Medicine, Rehabilitation and Occupational Medicine at the Medical University of Vienna
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
anxiety, depression, stress: HADS-D | 5 minutes
  HADS-D is a validated screening tool (questionnaire) to assess anxiety and depression in patients with physical and psychological disorders, especially taking into account a physical primary disease.

SECONDARY OUTCOMES:
anthropometric data (weight, height, body mass index) | 3 minutes
  weight, height and body mass index are measured
Psycho-oncologic basis assessment (PO-BADO) | 25-30 minutes
  The PO-BADO is a rating scale to assess the subjectively perceived stress in oncologic patients. The assessment is performed by a physician. Sociodemographic and medical data as well as psychologic distress are evaluated. Further relevant sociodemographic and medical data is assessed by a physician.
Visual analog scale (VAS) | 2 minutes
  The visual analog scale is a semiquantitative test to assess subjective pain intensity on a scale between 0-10 (0 being no pain at all, 10 being the worst pain imaginable). The patient is asked to report the most intense pain within the last week that is associated with the cancer diagnosis/treatment as well as musculoskeletal pain.
functional assessment: hand grip strength | 5 minutes
  Hand grip strength measures the maximal isometric handgrip strength using a JAMAR®dynamometer (in kilograms). Assessment is performed in a standardized position, sitting on a chair, elbow is flexed 90 degrees, upper extremity is in neutral position. 3 assessments are performed with the dominant hand, the mean value is registered. The motoric skill strength is assessed.
functional assessment: 6 Minute Walking Test | 8 minutes
  The 6 Minute Walking Test (6MWT) is used to estimate the basic motoric function endurance. It helps to evaluate the patients cardiovascular and pulmonal performance below the anerobic threshold. The patient is asked to quickly walk (not run) for 6 minutes, the distance walked within 6 minutes is measured. Walking aids and taking a break if needed is allowed. This test has been validated and recommended for cancer patients.
functional assessment: Timed Get up and Go Test | 5 minutes
  Timed Get up and Go Test (TGU): this standardized test assesses functional mobility. The patient is asked to sit on a chair with armrests. When told, he has to get up without the help of other persons, walk a distance of 3 meters, turn and sit down again. Walking aids such as a cane are allowed to use if necessary. The time is registered that the person needs for that maneuver (< 10 seconds indicate no limitations in mobility). The test has a good validity and reliability.
Quality of life: Short- Form -36 | 10 minutes
  The Short Form -36 is a validated questionnaire to assess the health-related quality of life. There are 8 dimensions of the test that can be summarized into the main domains "physical health" and "mental health". Also, changes compared to the year before are evaluated.
subjective perceived stress: Perceived Stress Scale (PSS-10) | 5 minutes
  The PSS-10 scale measures the subjective perception of stress. 2 scales evaluate the domains "helplessness" and "self-efficacy".
resilience: resilience scale (RS-13) | 5 minutes
  Resilience is seen as a criterion of emotional stability and psychological health. It is a personal resource to deal with stressful events in life. This one-dimensional scale evaluates the resilience of a person.
fatigue: brief fatigue inventory (BFI) | 5 minutes
  The BFI score is a validated tool to assess cancer-related fatigue. The questionnaire consists of 10 items that capture 6 dimensions: activity, mood, mobility, work, social relation and vitality.
disability related to pain: Pain Disability Index (PDI) | 5 minutes
  The PDI is used to assess the subjective impairment of a chronic pain situation in everyday life. The questionnaire is based on a multidimensional concept of impairment due to the pain condition. It differentiates between damage, disability and discrimination. It evaluates 7 areas of life (family/home, recreation, social activities, work, sexuality, self-supply, vital activities.)
workability: Work Ability Index - short version (WAI-K) | 5 minutes
  The WAI evaluates the amount to which employed people are able to do their work in light of health, mental resources and work requirements. It helps to estimate the individual performance regarding the current working situation. It consists of 10 items and 7 dimensions. The summary score is a measure for the subjective estimate of the own capacity to meet work requirements.
psychological assessment according to the diagnostic I.C.D.-10 based checklists | 90 minutes
  The psychological assessment is based on the results of the screening tools to identify psychosocial stress/ disorders. It aims to further evaluate the present problems and clarify whether symptoms are subsyndromal or fulfil the criteria of a mental disorder according to the I.C.D.-10 classification. External assessment tools used are the international diagnostic checklist for I.C.D.-10 (IDCL) and the I.C.D.-10 symptom checklist for mental disorders (SCL).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Crevenna, Prof MD MBA MMSc, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehnert A, Koch U. Psychosocial care of cancer patients--international differences in definition, healthcare structures, and therapeutic approaches. Support Care Cancer. 2005 Aug;13(8):579-88. doi: 10.1007/s00520-005-0779-6. Epub 2005 Mar 1. PMID 15739056
- [Background] Mehnert A, Lehmann C, Cao P, Koch U. [Assessment of psychosocial distress and resources in oncology--a literature review about screening measures and current developments]. Psychother Psychosom Med Psychol. 2006 Dec;56(12):462-79. doi: 10.1055/s-2006-951828. German. PMID 17160791
- [Background] Fallowfield L, Ratcliffe D, Jenkins V, Saul J. Psychiatric morbidity and its recognition by doctors in patients with cancer. Br J Cancer. 2001 Apr 20;84(8):1011-5. doi: 10.1054/bjoc.2001.1724. PMID 11308246
- [Background] Herschbach P, Book K, Brandl T, Keller M, Lindena G, Neuwohner K, Marten-Mittag B. Psychological distress in cancer patients assessed with an expert rating scale. Br J Cancer. 2008 Jul 8;99(1):37-43. doi: 10.1038/sj.bjc.6604420. Epub 2008 Jun 24. PMID 18577997
- [Background] Herschbach P, Keller M, Knight L, Brandl T, Huber B, Henrich G, Marten-Mittag B. Psychological problems of cancer patients: a cancer distress screening with a cancer-specific questionnaire. Br J Cancer. 2004 Aug 2;91(3):504-11. doi: 10.1038/sj.bjc.6601986. PMID 15238979
- [Background] Harkonen R, Harju R, Alaranta H. Accuracy of the Jamar dynamometer. J Hand Ther. 1993 Oct-Dec;6(4):259-62. doi: 10.1016/s0894-1130(12)80326-7. PMID 8124439
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Casanova C, Celli BR, Barria P, Casas A, Cote C, de Torres JP, Jardim J, Lopez MV, Marin JM, Montes de Oca M, Pinto-Plata V, Aguirre-Jaime A; Six Minute Walk Distance Project (ALAT). The 6-min walk distance in healthy subjects: reference standards from seven countries. Eur Respir J. 2011 Jan;37(1):150-6. doi: 10.1183/09031936.00194909. Epub 2010 Jun 4. PMID 20525717
- [Background] Manttari A, Suni J, Sievanen H, Husu P, Vaha-Ypya H, Valkeinen H, Tokola K, Vasankari T. Six-minute walk test: a tool for predicting maximal aerobic power (VO2 max) in healthy adults. Clin Physiol Funct Imaging. 2018 May 31. doi: 10.1111/cpf.12525. Online ahead of print. PMID 29851229
- [Background] Schmidt K, Vogt L, Thiel C, Jager E, Banzer W. Validity of the six-minute walk test in cancer patients. Int J Sports Med. 2013 Jul;34(7):631-6. doi: 10.1055/s-0032-1323746. Epub 2013 Feb 26. PMID 23444095
- [Background] Klein EM, Brahler E, Dreier M, Reinecke L, Muller KW, Schmutzer G, Wolfling K, Beutel ME. The German version of the Perceived Stress Scale - psychometric characteristics in a representative German community sample. BMC Psychiatry. 2016 May 23;16:159. doi: 10.1186/s12888-016-0875-9. PMID 27216151
- [Background] Radbruch L, Sabatowski R, Elsner F, Everts J, Mendoza T, Cleeland C. Validation of the German version of the brief fatigue inventory. J Pain Symptom Manage. 2003 May;25(5):449-58. doi: 10.1016/s0885-3924(03)00073-3. PMID 12727043
- [Background] van den Berg TI, Elders LA, de Zwart BC, Burdorf A. The effects of work-related and individual factors on the Work Ability Index: a systematic review. Occup Environ Med. 2009 Apr;66(4):211-20. doi: 10.1136/oem.2008.039883. Epub 2008 Nov 18. PMID 19017690